CLINICAL TRIAL: NCT00759512
Title: Effects of Therapeutic Touch on Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Ann Smith, PhD, University of Toledo, Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UTHSC - 09
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Osteoarthritis in the Knee
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): This arm received the Kreiger/Kunz method of Therapeutic Touch in addition to Standard of Care
  Interventions: Other: Therapeutic Touch
- Arm 2 (No Intervention): Standard of Care

INTERVENTIONS:
Other: Therapeutic Touch
  Arms: Arm 1

SUMMARY:
This study is to evaluate the efficacy of the Kreiger/Kunz method of Therapeutic Touch on function, pain perception and quality of life in persons with Osteoarthritis in the knee.

ELIGIBILITY:
Inclusion Criteria:

* Persons diagnosed with or exhibiting signs of osteoarthritis of at least one knee.

Exclusion Criteria:

* Persons with connective tissue disorder
* Persons with bilateral total joint replacement of the knee
* Persons with dementia
* Persons with a systemic illness producing joint symptoms

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-08; Primary Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
SF36 | 8, 12, 16 weeks
WOMAC | 8, 12 and 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ann Smith, PhD, Principal Investigator — UT, Health Science Campus
Locations (1):
- University of Toledo, Health Science Campus, Toledo, Ohio, United States